CLINICAL TRIAL: NCT00282802
Title: Twins and the Risk of PD: A Clinical and Imaging Study
Brief Title: Twins and the Risk of Parkinson's Disease: A Clinical and Imaging Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Parkinson's Institute (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Caroline M. Tanner, MD, PhD, Director of Clinical Research, The Parkinson's Institute
Other Study IDs: R01NS040467 (NIH); R01NS040467-01 (NIH)
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; twins; SPECT; National Academy of Sciences/National Resource Council (NAS/NRC) World War II Veteran Twins Cohort Registry; NAS/NRC; World War II Veteran Twins
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: National Academy of Sciences/National Resource Council (NAS/NRC) World War II Veteran Twins Cohort

SUMMARY:
The purpose of this study is to examine the role of genetic and environmental factors in the cause of Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a growing health problem in the elderly, and genetic factors may provide substantial clues toward eventual treatment and/or prevention of the disorder. The National Academy of Sciences/National Resource Council (NAS/NRC) World War II (WWII) Veteran Twins Cohort Registry is one of the few population-based groups of elderly twins. Previous studies in this group indicated that genetic factors were involved only in early-onset PD, however there was no follow-up to these studies.

The purpose of the "Twins and the Risk of PD" study is to follow-up previous studies and confirm the initial findings. In this study, investigators will use the NAS/NRC WWII Veteran Twin Cohort Registry to compare the concordance rates for PD in monozygotic and dizygotic twins-at least one of whom has PD.

The overall goal of this research is determine the contributions of genetic and environmental factors in the cause of PD.

The study will involve traditional clinical research methods, such as a clinical examination, as well as innovative imaging techniques, such as single photon emission computed tomography (SPECT). SPECT-a nuclear imaging test involving blood flow to tissue-is used to evaluate certain brain functions.

Findings from this study may help to set research priorities in PD, and to develop tools for early detection of the disorder.

ELIGIBILITY:
Inclusion:

* Participants will be recruited from a closed cohort-the National Academy of Sciences/National Resource Council (NAS/NRC) World War II Veteran Twins Cohort

Ages: 77 Years to 88 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants will be recruited from a closed cohort-the National Academy of Sciences/National Resource Council (NAS/NRC) World War II Veteran Twins Cohort
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2001-04; Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Onset of Parkinson's disease | duration of the project

SECONDARY OUTCOMES:
Age of Parkinson's disease onset | duration of the project

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M. Tanner, MD, Principal Investigator — The Parkinson's Institute
Locations (1):
- The Parkinson's Institute, 675 Almanor Avene, Sunnyvale, California, United States